CLINICAL TRIAL: NCT02815137
Title: Prevalence, Kinetic and Prognostic Value of XPO1 E571K Mutation Detection in Plasma Cell-free DNA From Patients Xith Classical Hodgkin Lymphoma
Brief Title: Detection and Prognostic Value of Recurrent XPO1 Mutations of Patients With Classical Hodgkin Lymphoma
Acronym: XPO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB 16.02
Record Dates: First submitted 2016-06-13; First posted 2016-06-28 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Digital PCR; classical; Hodgkin Lymphoma; mutation
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XPO1 E571K mutation detection (Other): Determination of mutation of XPO1571K in patient with classical hodgkin Lymphoma by digital PCR on blood samples and biopsy
  Interventions: Other: Digital Polymerase Chain Reaction

INTERVENTIONS:
Other: Digital Polymerase Chain Reaction — Determination of mutation of XPO1 E571K by digital PCR in blod sample of patient with classical hodgkin lymphoma

SUMMARY:
The purpose of this study is to determine if the XPO1 E571K mutation could be used as molecular residual disease biomarker in classical Hodgkin's lymphoma. To determine the interest of the mutation assessment by digital Polymerase Chain Reaction, sensitivity and specificity after 2 courses of chemotherapy (C2) will be compared with the deltaSUVmax determined by Positron Emission Tomography after C2 and at end of treatment.

DETAILED DESCRIPTION:
A research team of Centre Henri Becquerel recently detected an unexpected recurrent point mutation of XPO1 (exportin 1) (also known as Chromosome Region Maintenance 1) located in exon 15 (c.1711G>A) leading to the Glu571Lys (p.E571K) missense substitution in relapsed/refractory (R/R) Primary Mediastinal Large B-cell Lymphoma (PMBL) patients included in the LYSA LNH03 trial program and in classical Hodgkin's Lymphoma patients. It was found recurrent XPO1 E571K mutations in a large cohort of 94 patients with classical Hodgkin's lymphoma. This observation is new and could add new information on driver events and tumorigenesis in this disease. In total, 24.2 % of the patients with classical Hodgkin's lymphoma harbored the XPO1 E571K mutation. It is remarkable that 29% of all XPO1 mutations were only found in the plasma but not in the tumor because of the well-known tumor cell sparsity in Hodgkin's lymphoma. In this particular disease, highly sensitive techniques like digital Polymerase Chain Reaction and targeted Next-Generation Sequencing are essential to highlight low frequency mutations. The research team of the Centre Henri Becquerel have identified a trend toward unfavorable prognostic impact in terms of progression-free survival in patients with detectable XPO1 E571K mutation in plasma cell-free DNA at the end of treatment, which could prove to be statistically significant in a larger cohort. It was observed that 57% of patients who ultimately relapsed were positive in the plasma after end of therapy. It remains to be established whether this mutation adds new relevant value as compared to Positron Emission Tomography-scan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Pathologically confirmed, recent diagnosis of classical Hodgkin Lymphoma
* treatment planned with Adriamycin Bleamycin Vinblastine Dacarbazine (ABVD) or Bleomycin Etoposide Adriamycin Cyclophosphamide Vincristine Procarbazine Prednisone (BEACOPP) regimen (and radiotherapy if applicable)
* all stages (Ann Arbor I - IV)
* Written informed consent
* Patient affiliated or beneficiary of a benefit system
* untreated patient (no corticosteroids or chemotherapy)

Exclusion Criteria:

* No informed consent
* Treatment by ABVD or BEACOPP not indicated
* Previously treated Hodgkin lymphoma (including corticosteroids)
* Patients who are pregnant or lactating
* Active Hepatitis B or Hepatitis C infection
* Known human immunodeficiency virus (HIV) infection - Patient with no social protection
* Patient under tutorship or curatorship
* Patient not affiliated of beneficiary of a benefit system
* Medical contraindication to PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
If the mutation can be used as a molecular minimal residual disease biomarker | 56 days
  Comparison of the sensitivity and specificity of the detection of the mutation between delta Standard Uptake Value max (SUV max) determined by PET after two courses of chemotherapy

SECONDARY OUTCOMES:
Kinetic of allele frequency decrease | 224 days
  difference between the variant allele fraction at the end of treatment and at the diagnosis
Variation of Deauville scale | 224 days
  Difference of metabolic parameter in TEP between the end of treatment and the diagnosis
Progression-free survival | 2 years
  Time between the inclusion and the date of progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice JARDIN, PUPH, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camus V, Viennot M, Lequesne J, Viailly PJ, Bohers E, Bessi L, Marcq B, Etancelin P, Dubois S, Picquenot JM, Veresezan EL, Cornic M, Burel L, Loret J, Becker S, Decazes P, Lenain P, Lepretre S, Lemasle E, Lanic H, Menard AL, Contentin N, Tilly H, Stamatoullas A, Jardin F. Targeted genotyping of circulating tumor DNA for classical Hodgkin lymphoma monitoring: a prospective study. Haematologica. 2021 Jan 1;106(1):154-162. doi: 10.3324/haematol.2019.237719. PMID 32079702